CLINICAL TRIAL: NCT04911062
Title: A Phase 2, Two-Part, Multicenter Study of HTX-011 in Spinal Surgery
Brief Title: HTX-011 in Spinal Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Heron Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HTX-011-221
Record Dates: First submitted 2021-05-27; First posted 2021-06-02 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-06

CONDITIONS: Post-Operative Pain; Lumbar Laminectomy
Keywords: postoperative pain; local anesthetic; lumbar laminectomy; lumbar decompression
MeSH Terms: conditions — Pain, Postoperative | interventions — Epinephrine

STUDY DESIGN:
Masking Description: Optional Part B will be randomized, blinded, active-controlled.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (3):
- Cohort 1: Bupivacaine HCl (Experimental): Bupivacaine HCl without epinephrine, via injection into the surgical site.
  Interventions: Drug: Bupivacaine HCI without epinephrine
- Cohort 2: HTX-011 (Experimental): HTX-011 (bupivacaine/meloxicam) via application into the surgical site.
  Interventions: Drug: HTX-011; Device: Luer Lock Applicator
- Cohort 3: HTX-011 (Experimental): HTX-011 (bupivacaine/meloxicam) via application into the surgical site.
  Interventions: Drug: HTX-011; Device: Luer Lock Applicator

INTERVENTIONS:
Drug: Bupivacaine HCI without epinephrine — 100 mg administered via injection into the surgical site.
  Arms: Cohort 1: Bupivacaine HCl
Drug: HTX-011 — HTX-011 (bupivacaine/meloxicam) dose up to 200 mg/6 mg administered via application into the surgical site.
  Arms: Cohort 2: HTX-011; Cohort 3: HTX-011
Device: Luer Lock Applicator — Applicator for instillation.
  Arms: Cohort 2: HTX-011; Cohort 3: HTX-011

SUMMARY:
This is a Phase 2, multicenter study in subjects undergoing an open lumbar decompression surgery.

ELIGIBILITY:
Inclusion Criteria:

* Is scheduled to undergo an open 1-3 level lumbar decompression surgery with or without fixation under general anesthesia.
* Females are eligible only if not pregnant, not lactating, not planning to become pregnant during the study.

Exclusion Criteria:

* Has a contraindication of a known or suspected history of hypersensitivity or clinically significant idiosyncratic reaction to required study medications.
* Has a history of severe allergic reaction due to aspirin or other NSAIDs, or known history of severe gastrointestinal adverse reactions associated with NSAID use.
* Has functioning intrathecal drug pump or spinal cord stimulator.
* Opioid use for most days within the last 3 months.
* Has initiated treatment with selective serotonin reuptake inhibitors (SSRIs), selective norepinephrine reuptake inhibitors (SNRIs), gabapentin, pregabalin, or duloxetine within 1 month prior to the scheduled surgery.
* Received an investigational product or device in a clinical trial within 30 days or within 5 elimination half-lives.
* Has a history of clinically significant cardiac abnormality, coronary artery bypass graft surgery within 12 months, or suspected coagulopathy or uncontrolled anticoagulation.
* Has impaired balance and is at risk of falling.
* Is currently undergoing treatment for hepatitis B, hepatitis C, or HIV.
* Has undergone 3 or more surgeries within 12 months.
* Has a known history of glucose-6-phosphate dehydrogenase deficiency.
* Has History of liver cirrhosis, having an aspartate aminotransferase >3 × the upper limit of normal (ULN), or having an alanine aminotransferase >3 × ULN.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2022-04-07 (Actual); Primary Completion 2022-07-29 (Actual); Study Completion 2022-08-26 (Actual)

PRIMARY OUTCOMES:
Incidence of Serious Adverse Events | From the time the subject signs the ICF through the Day 29 Visit

SECONDARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) | Baseline through 120 hours
Time of occurrence of maximum concentration (Tmax) | Baseline through 120 hours
Area under the concentration-time curve from Time 0 to the time of last quantitative concentration (AUClast) | Baseline through 120 hours
Area under the concentration-time curve from Time 0 extrapolated to infinity (AUCinf) | Baseline through 120 hours
Apparent terminal half-life (t½) | Baseline through 120 hours

CONTACTS AND LOCATIONS:
Locations (12):
- United States (12):
  - Arizona Research Center, Phoenix, Arizona
  - Lotus Clinical Research, LLC, Pasadena, California
  - Kansas Spine and Specialty Hospital, Wichita, Kansas
  - Spine Institute of Louisiana, Shreveport, Louisiana
  - Overlook Medical Center, Summit, New Jersey
  - M3 Emerging Medical Research, LLC, Durham, North Carolina
  - The Ohio State University Wexner Medical Center - University Hospital, Columbus, Ohio
  - Austin Neurosurgeons, Austin, Texas
  - First Surgical Hospital, Bellaire, Texas
  - Houston Heights Hospital, Houston, Texas
  - South Texas Spine & Surgical Center, San Antonio, Texas
  - JBR Clinical Research, Salt Lake City, Utah